CLINICAL TRIAL: NCT05583019
Title: Device Quantification of Scratch and Sleep in Atopic Dermatitis With Accelerometry and Polysomnography (ADAP) Study
Brief Title: Atopic Dermatitis With Accelerometry and Polysomnography (ADAP)
Acronym: ADAP
Status: Completed | Type: Observational
Sponsor: SymmetryScience Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SSG0001
Record Dates: First submitted 2022-10-14; First posted 2022-10-17 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis; Eczema; Healthy
Keywords: Atopic Dermatitis; Eczema; Healthy
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Control: Those who do not have a diagnosis of Atopic Dermatitis (AD) or eczema and score a Clear (0) or Almost Clear (1) on the Investigator's Static Global Assessment (ISGA) at intake.
  Interventions: Device: GENEActiv Accelerometry Device; Device: Centrepoint Insights Watch (CPIW) Accelerometry Device; Device: Apple Watch Accelerometry Device; Device: Polysomnography; Device: Videography
- Mild Atopic Dermatitis (AD): Those who have a diagnosis of Atopic Dermatitis (AD) or eczema and score a Mild (2) on the Investigator's Static Global Assessment (ISGA) at intake.
  Interventions: Device: GENEActiv Accelerometry Device; Device: Centrepoint Insights Watch (CPIW) Accelerometry Device; Device: Apple Watch Accelerometry Device; Device: Polysomnography; Device: Videography
- Moderate Atopic Dermatitis (AD): Those who have a diagnosis of Atopic Dermatitis (AD) or eczema and score a Moderate (3) on the Investigator's Static Global Assessment (ISGA) at intake.
  Interventions: Device: GENEActiv Accelerometry Device; Device: Centrepoint Insights Watch (CPIW) Accelerometry Device; Device: Apple Watch Accelerometry Device; Device: Polysomnography; Device: Videography
- Severe Atopic Dermatitis (AD): Those who have a diagnosis of Atopic Dermatitis (AD) or eczema and score a Severe (4) on the Investigator's Static Global Assessment (ISGA) at intake.
  Interventions: Device: GENEActiv Accelerometry Device; Device: Centrepoint Insights Watch (CPIW) Accelerometry Device; Device: Apple Watch Accelerometry Device; Device: Polysomnography; Device: Videography

INTERVENTIONS:
Device: GENEActiv Accelerometry Device — a watch like wearable sensor
  Other Names: GENEActiv Watch
Device: Centrepoint Insights Watch (CPIW) Accelerometry Device — a watch like wearable sensor
  Other Names: Centrepoint Insights Watch (CPIW)
Device: Apple Watch Accelerometry Device — a watch like wearable sensor
  Other Names: Apple Watch
Device: Polysomnography — Sleep monitor
Device: Videography — Thermal Camera

SUMMARY:
The purpose of this research is to better understand how wrist-worn study devices that measure activity/motion ('accelerometry devices') can be used to assess scratching and sleep in participants aged 12-75 years, with and without Atopic Dermatitis (AD, eczema), in both a sleep laboratory (hotel) setting and in a daily life/home setting. In this study, we will be using three different wrist devices to collect information: an Apple Watch Series 7, an Actigraph CentrePoint Insights Watch (CPIW) and a GENEActiv Original Watch. We will also compare the movement and sleep measurements recorded on the devices to thermal video and sleep assessments done in the sleep laboratory (hotel) as well as compare them to Patient Reported Outcome (PRO) assessments.

DETAILED DESCRIPTION:
The general procedures include an initial intake appointment on day 1 (can be completed up to 3 days prior in case of scheduling conflicts), two overnight sleep laboratory visits, followed by approximately 12 days of wearing the devices during the participant's normal day-to-day activities and answering questions on a study-provided iPhone in the routine/home setting. The participant will be asked to complete questionnaires related to itch, sleep, pain, and overall Atopic Dermatitis (AD) severity each day, as relevant, and continuously wear wrist-worn accelerometry devices (as specified) during the study.

The study will begin with an initial in-laboratory intake appointment to verify study eligibility to participate in the study. We do our best to screen for study eligibility over the phone, but there are some eligibility requirements that must be assessed in person. This means that at the first appointment, there is a chance that the prospective participant will not be eligible to continue with the remainder of study activities. In the event that they are not eligible to continue at the first in- person appointment, they will be compensated a prorated study amount for their time.

Following the initial intake appointment, the participant will sleep overnight at the sleep laboratory/hotel. The participant will wear both the Apple Watch and the CentrePoint Insights Watch (CPIW) wrist devices, one of each, on both wrists. They will be asked to don the devices at least 6 hours before bedtime on the first overnight visit (day 1) and wear devices continuously (as specified) thereafter. The participant will be video recorded with an infra-red thermal camera (this video is de-identified, and only shows a heat map of their body, so facial features cannot be seen) during the sleep laboratory/hotel visits, wear the wrist accelerometry devices, and complete electronic questionnaires. In addition, on the second overnight in the sleep lab they will also have sensors placed on their head and limbs to monitor their sleep. Both nights, all three devices will also be next to the participant on the night stand, collecting information about their surroundings while they sleep. Upon the completion of the second night in the sleep laboratory (Days 1 and 2), they will then continue to wear wrist accelerometry devices and complete Patient Reported Outcome (PRO) questionnaires at home. The participants will be split into two cohorts (groups): Cohort 1 will wear both the CPIW and the GENEActiv device on both wrists and Cohort 2 will wear both the Apple Watch and GENEActiv device on both wrists. The participants will return to the laboratory on day 8 (+/- 2 days) to swap out devices. Cohort 1 will then wear both the Apple Watch and the GENEActiv device on both wrists and Cohort 2 will wear both the CPIW and GENEActiv device on both wrists for the remaining study days. At the conclusion of the at-home portion of the study, the participant will return the devices and assessments to the laboratory and complete final assessments.

ELIGIBILITY:
Inclusion Criteria:

Atopic Dermatitis (AD) Participants:

1. Participants aged ≥12 years of age and <75 years of age at Day 1.
2. Written informed consent from participant or parent(s)/guardian(s) and assent from the participant (where assent is applicable).
3. Participant (and parent(s)/guardian(s)) are willing and able to comply with study instructions, study visits, and procedures.
4. Native English speakers or demonstrated fluency in English (participant; and parent(s)/guardian(s) as needed)
5. Have a clinical diagnosis of AD according to the criteria of Hanifin and Rajka (concomitant AD treatments are permitted on study).
6. Have AD involvement ≥ 5% Treatable % Body Surface Area (BSA) excluding the scalp.
7. Have an Investigator's Static Global Assessment (ISGA) score of Mild (2), Moderate (3) or Severe (4) at the screening visit within 14 days of study enrollment.
8. Have a minimum Peak Pruritus Numerical Rating Scale (PP-NRS) assessment score of 3 (out of 10).
9. Wide Range Achievement Test-4 (WRAT-4) Word Reading Subtest equivalent to 8th grade reading level or greater (for ages ≥18 years only).

Healthy (non-AD) Participants:

1. Participants aged ≥12 years of age and <75 years of age at Day 1.
2. Written informed consent from participant or parent(s)/guardian(s) and assent from the participant (where assent is applicable).
3. Participant (and parent(s)/guardian(s)) are willing and able to comply with study instructions, study visits, and procedures.
4. Native English speakers or demonstrated fluency in English (participant; and parent(s)/guardian(s) as needed)
5. Does not have suspected or confirmed clinical diagnosis of AD (according to the criteria of Hanifin and Rajka).
6. Have an ISGA score of Clear (0) or Almost Clear (1) at the screening visit within 14 days of study enrollment.
7. WRAT-4 Word Reading Subtest equivalent to 8th grade reading level or greater (for ages ≥18 years only).

Exclusion Criteria:

Atopic Dermatitis (AD) Participants:

1. Has any clinically significant medical disorder, condition, disease (including active or potentially recurrent non-AD dermatological conditions and known genetic dermatological conditions that overlap with AD, such as Netherton syndrome) or clinically significant finding at screening that precludes participant's participation in study activities.
2. Allergy to polyurethane resin (strap/wristband component).
3. Has documented non-AD related insomnia, sleep apnea or other sleep-related disorders (e.g., narcolepsy, restless legs syndrome, circadian rhythm disorder).
4. AD affected surface areas are in a location of device placement.
5. If participant has a history of angioedema or anaphylaxis and has had any anaphylactic reactions within the past 6 months.
6. Has unstable AD (Total BSA>40%).
7. Has a significant active systemic or localized infection, including actively infected AD.
8. Has recently (within 30 days of Day 1) participated in or is currently involved in another drug or device research study for AD.
9. Has any planned surgical or medical procedure that would overlap with study participation.
10. Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are employees directly involved in the conduct of the study.
11. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) wine, 12 ounces (360 mL) of beer, or 1.5 ounces (45 mL) of hard liquor) within 6 months of baseline as disclosed by participant during evaluation (for those participants over the age of 21).
12. Is a female who is breastfeeding or pregnant, as disclosed by the participant.
13. Current shift worker or travel across more than two time zones in the past 2 weeks, and/or during the study period.
14. Participants with cardiac pacemakers, electronic pumps or any other implanted medical devices.

Healthy (non-AD) Participants:

1. Has any clinically significant medical disorder, condition, disease (including any active/potentially recurrent dermatological conditions (such as Netherton syndrome) or clinically significant finding at screening that precludes participant's participation in study activities.
2. Allergy to polyurethane resin (strap/wristband component).
3. Has documented clinically diagnosed insomnia, sleep apnea or other sleep-related disorders (e.g., narcolepsy, restless legs syndrome, circadian rhythm disorder).
4. If participant has a history of angioedema or anaphylaxis and has had any anaphylactic reactions within the past 6 months.
5. Has recently (within 30 days of Day 1) participated in or is currently involved in another drug or device research study.
6. Has any planned surgical or medical procedure that would overlap with study participation.
7. Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are employees directly involved in the conduct of the study.
8. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) wine, 12 ounces (360 mL) of beer, or 1.5 ounces (45 mL) of hard liquor) within 6 months of baseline as disclosed by participant during evaluation (for those participants over the age of 21).
9. Is a female who is breastfeeding or pregnant, as disclosed by the participant.
10. Current shift worker or travel across more than two time zones in the past 2 weeks, and/or during the study period.
11. Participants with cardiac pacemakers, electronic pumps or any other implanted medical devices.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Participants over or including the age of 12 and under the age of 75 Participants with Atopic Dermatitis (AD) over or including the age of 12 and under the age of 75
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Quantification of scratch using GENEActiv watches to assess triaxial accelerometry | 14 days +/- 2 days
  One GENEActiv watch will be used on each wrist at a sampling rate of 100 Hz to measure movement in the x, y, and z direction.
Quantification of scratch using Centrepoint Insights Watches (CPIW) to assess triaxial accelerometry | 14 days +/- 2 days
  One CPIW watch will be used on each wrist at a sampling rate of 128 Hz to measure movement in the x, y, and z direction.
Quantification of scratch using Apple Watches to assess triaxial accelerometry | 14 days +/- 2 days
  One Apple Watch will be used on each wrist at a sampling rate of 100 Hz to measure movement in the x, y, and z direction.
Quantification of sleep occurrences using polysomnography | 1 night
  Polysomnography (PSG) will be used to report the number of sleep occurrences based on the scoring guide provided by the American Academy of Sleep Medicine (AASM).
Sleep stage scoring using polysomnography | 1 night
  Polysomnography (PSG) will be used to report the appropriate sleep staging based on the scoring guide provided by the American Academy of Sleep Medicine (AASM). The following sleep stages will be scored: Stage W (wakefulness), Stage N1 (NREM 1), Stage N2 (NREM 2), Stage N3 (NREM 3), Stage N (NREM), and Stage R (REM).

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Moss, PhD, Principal Investigator — SymmetryScience Group, Inc.
Locations (1):
- Hampton Inn & Suites, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No